CLINICAL TRIAL: NCT02944253
Title: Ketosis and Appetite Suppression - What is the Maximum Carbohydrate Intake That is Still Associated With Appetite Suppression in a Low Energy Diet?
Brief Title: What is the Maximum Amount of Carbohydrates That is Still Able to Induce Ketosis and Suppress Appetite?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/1297
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: Diet, Reducing; Hunger; Appetite Regulation; Ketogenic Diet; Caloric Restriction; Weight Loss; Ketosis
MeSH Terms: conditions — Obesity; Weight Loss; Ketosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low energy diet 70 gram carbohydrates (Experimental): isocaloric 4128 kilojoules/day (1000 kilocalories/day) for men and women, low energy diet containing 70 gram carbohydrates for 8 weeks.
  Interventions: Other: Low energy diet 70 gram carbohydrates
- Low energy diet 100 gram carbohydrates (Experimental): isocaloric (4128 kilojoules/day (1000 kilocalories/day) for men and women, low energy diet containing 100 gram carbohydrates for 8 weeks.
  Interventions: Other: Low energy diet 100 gram carbohydrates
- Low energy diet 130 gram carbohydrates (Experimental): isocaloric 4128 kilojoules/day (1000 kilocalories/day) for men and women, low energy diet containing 130 gram carbohydrates for 8 weeks.
  Interventions: Other: Low energy diet 130 gram carbohydrates

INTERVENTIONS:
Other: Low energy diet 70 gram carbohydrates — isocaloric 4128 kilojoules/day (1000 kilocalories/day) for men and women, low energy diet containing 70 gram carbohydrates
  Arms: Low energy diet 70 gram carbohydrates
Other: Low energy diet 100 gram carbohydrates — isocaloric 4128 kilojoules/day (1000 kilocalories/day) for men and women
  Arms: Low energy diet 100 gram carbohydrates
Other: Low energy diet 130 gram carbohydrates — isocaloric 4128 kilojoules/day (1000 kilocalories/day) for men and women, low energy diet containing 130 gram carbohydrates
  Arms: Low energy diet 130 gram carbohydrates

SUMMARY:
Two dietary approaches, very low energy diets (VLEDs) and ketogenic low carbohydrate diets (KLCDs), have the ability to suppress appetite. The suppression of appetite typically observed during these diets is believed (but not clinically proven) to be due to ketosis, a condition where circulating concentrations of ketone bodies are increased due to a higher production of ketones in the liver. Little is known about the potential mechanisms through which ketosis may lead to appetite suppression in VLEDs and KLCDs. A 'ketogenic diet' typically contains less than 50 grams carbohydrate per day, yet ketosis has been seen in subjects who consume diets with a carbohydrates ranging between 59-192 grams per day. Although an association between ketosis and appetite suppression has been established, the minimum level of ketosis and maximum carbohydrate intake that is still associated with appetite suppression remains unknown and should be explored. The ability to increase carbohydrate intake while maintaining a suppressed appetite will allow dieters to consume more carbohydrate-rich food that is beneficial for health without feeling more hungry.

The study, 'can Appetite Suppression be achieved using KEtogenic Diets with more carbohydrates?' (ASKED) aimed to:

* to identify the maximum carbohydrate intake that is still associated with appetite suppression in a low energy diet and to determine the impact of a higher carbohydrate intake on appetite suppression, ketosis, body composition, and resting metabolic rate. A
* to evaluate the impact of weight loss while in and out of ketosis on markers of appetite (appetite related hormones and appetite sensations measured using visual analogue scales).

DETAILED DESCRIPTION:
A total of 101 healthy, weight stable (< 2 kg variation in BW within the last 3 months), adult (18-65 years old) individuals with obesity (body mass index [BMI] 30-45 kg/m2) who were not actively trying to lose weight were recruited through advertisements in Facebook, Twitter and the intranet of St. Olavs Hospital and the Norwegian University of Science and Technology (NTNU) in Trondheim, Norway from May 2017 - August 2018.

Informed consent was obtained from all participants before enrollment in the study, and participants were allowed to withdraw at any time.

Study participants were randomized to one of three intervention arms: low, medium, or high CHO groups. Computer-generated randomization was performed using a block sampling (fixed block size) and stratification approach to account for the potential confounding factors of sex and BMI (< 35 and ≥ 35 kg/m2). (34, 35). Study participants were not made aware of which intervention arm they were allocated to until the end of the trial. All participants underwent an 8-week, supervised LED containing different amounts of CHO, followed by 4 weeks of gradual refeeding and weight stabilization. Measurements were taken before diet initiation (baseline), at the end of the WL phase (week 8) and at the end of the weight stabilization phase (week 12) to allow for the evaluation of the impact of WL in or out of ketosis on appetite markers.

ELIGIBILITY:
Inclusion Criteria:

* class I or II obesity (BMI 30-45 kg/m2)
* weight stable (<2 kg variation in weight within the last 3 months)
* not currently dieting to lose weight
* women who are either post-menopausal, taking oral contraceptives or with a normal cycle (28 ± 2 days)

Exclusion Criteria:

* pregnant
* breast-feeding
* drug or alcohol abuse within the last two years
* currently taking medication known to affect appetite or induce weight loss
* enrolled in another obesity treatment program
* history of psychological disorders
* having had bariatric surgery
* metabolic diseases (such as hypo/hyperthyroidism and diabetes type 1 or 2)
* eating disorders
* lactose intolerance
* gastrointestinal (particularly cholelithiasis), kidney, liver, lung, cardiovascular disease
* malignancies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Suppression of appetite sensations measured using online visual analogue scales | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Assessed by an online version of Visual Analogue Scale (VAS), a validated scale used to measure appetite sensations in response to questions posed regarding feelings of hunger, fullness, desire to eat, prospective consumption. Study participants are asked questions such as 'How hungry do you feel right now?' and are asked to provide a response by marking across a 100 millimeter long line with sentences anchored at each end such as "I have never been more hungry/ or I am not hungry at all" corresponding to their feeling. VAS measurements are done in fasting, immediately after a meal and every 30 minutes for 2.5 hours. Measurements are quantified by measuring the distance from the left end of the line to the mark indicated by the participant.
Suppression of appetite indicated by appetite-related hormones Active Ghrelin, Total Glucagon Like Peptide-1, Total Peptide YY and Insulin | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Measurement of plasma samples of appetite related hormones: Active ghrelin (AG), Total Glucagon Like Peptide-1 (Total GLP-1), Total Peptide YY (Total PYY) and Insulin measured in fasting, immediately after a meal and every 30 minutes for a period of 2.5 hours. Blood samples are first collected in Ethylenediaminetetraacetic acid (EDTA) tubes (72 milliliters in total) and centrifuged for 10 minutes at 18 degrees celsius with 3200 revolutions per minute (RPM). Plasma samples are then stored in -80 degree celsius freezer until analysis using a Metabolic Hormone Magnetic Bead Panel (Lincoplex Kit, Merck Millipore, USA). Results of plasma samples of these hormones will be presented in picograms (pg) per milliliter (ml).
Suppression of appetite indicated by appetite-related hormone Cholecystokinin (CCK) | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Measurement of plasma samples of appetite related hormone Cholecystokinin (CCK) measured in fasting, immediately after a meal and every 30 minutes for a period of 2.5 hours. Blood samples are first collected in Ethylenediaminetetraacetic acid (EDTA) tubes (72 milliliters in total inclusive of blood collected for analysis of hormones listed above) and centrifuged for 10 minutes at 18 degrees celsius with 3200 revolutions per minute (RPM). Plasma samples are then stored in -80 degree celsius freezer until they are sent to the University of Copenhagen to be analyzed by the research group of Professor Jens F Rehfeld using his 'In-house Radioimmunoassay method'. The results of plasma CCK will be presented in picomoles (pmol) per liter (l).
Ketosis | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period
  Measured with beta hydroxybutyrate (BHB), a ketone body and indicator of ketosis in plasma form. Fasting blood samples are first collected in Ethylenediaminetetraacetic acid (EDTA) tubes (inclusive of the 72 milliliters of blood collected for analysis of appetite hormones listed above) and centrifuged for 10 minutes at 18 degrees celsius with 3200 revolutions per minute (RPM). Plasma samples are then stored in -80 degree celsius freezer until analysis using a Ketone Body Assay (MAK-134, Merck Millipore, USA). The results of plasma BHB will be presented in millimoles (mmol) per liter (l).

SECONDARY OUTCOMES:
Body composition (air displacement plethysmography) | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Body composition measured with air displacement plethysmography (BodPod, COSMED, Italy). The output of the measurement of body composition using air displacement plethysmography provides absolute values in kilograms for body weight, fat mass and fat free mass.
Percent fat/fat-free mass (air displacement plethysmography) | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Percent fat mass and fat free mass is measured with air displacement plethysmography (BodPod, COSMED, Italy). The output of the measurement of body composition using air displacement plethysmography provides fat mass and fat free mass as a percentage of total body weight.
Body composition (bioelectrical impedance) | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Body composition measured using bioelectrical impedance analysis (BIA, Biospace, Korea). The output of the measurement of body composition using bioelectrical impedance analysis provides absolute values in kilograms for body weight, fat mass and fat free mass.
Percent fat/fat-free mass (bioelectrical impedance analysis) | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Percent fat mass and fat free mass is measured with bioelectrical impedance analysis (BIA, Biospace, Korea). The output of the measurement of body composition using bioelectrical impedance analysis provides fat mass and fat free mass as a percentage of total body weight.
Intracellular and extracellular water measured using Bioelectrical impedance analysis | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Intracellular and extracellular water is measured with bioelectrical impedance analysis (BIA, Biospace, Korea). The output of the measurement of body composition using bioelectrical impedance analysis provides information on the amount total body water (made up of intracellular and extracellular water) in liters.
Waist and hip circumference | 12 weeks (at start of study (baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Waist and hip circumference will be measured with a measuring tape and the results will be provided in centimeters.
Height | 12 weeks (at start of study (Baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Height of the participant will be measured with a stadiometer and will be provided in meters.
Body mass index (BMI) | 12 weeks (at start of study (Baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Body mass index (BMI) will be calculated using the measurements of body weight (obtained using the weight in kilograms output provided by bioelectrical impedance analysis) and height in meters measured using the stadiometer using the following formula: (kilograms/meters)^2
Resting metabolic rate | 12 weeks (at start of study (Baseline), at week 9 (after diet induced weight loss period), and week 13 (after weight stabilization period)
  Measured through indirect calorimetry. Indirect calorimetry is a technique that measures oxygen consumption and carbon dioxide production during rest to estimate resting metabolic rate. Results will be presented in kilocalories per day.

CONTACTS AND LOCATIONS:
Overall Officials: Magne Børset, phd prof, Study Chair — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deemer SE, Plaisance EP, Martins C. Impact of ketosis on appetite regulation-a review. Nutr Res. 2020 May;77:1-11. doi: 10.1016/j.nutres.2020.02.010. Epub 2020 Feb 20. PMID 32193016
- [Result] Martins C, Roekenes J, Salamati S, Gower BA, Hunter GR. Metabolic adaptation is an illusion, only present when participants are in negative energy balance. Am J Clin Nutr. 2020 Nov 11;112(5):1212-1218. doi: 10.1093/ajcn/nqaa220. PMID 32844188
- [Result] Martins C, Roekenes J, Gower BA, Hunter GR. Metabolic adaptation is associated with less weight and fat mass loss in response to low-energy diets. Nutr Metab (Lond). 2021 Jun 11;18(1):60. doi: 10.1186/s12986-021-00587-8. PMID 34116675
- [Result] Martins C, Nymo S, Aukan MI, Roekenes JA, Coutinho SR, Hunter GR, Gower BA. Association between ss-Hydroxybutyrate Plasma Concentrations after Hypocaloric Ketogenic Diets and Changes in Body Composition. J Nutr. 2023 Jul;153(7):1944-1949. doi: 10.1016/j.tjnut.2023.05.010. Epub 2023 May 12. PMID 37182692
- [Result] Martins C, Roekenes J, Salamati S, Gower BA, Hunter GR. Reply to E Ravussin and L Redman. Am J Clin Nutr. 2020 Dec 10;112(6):1655-1656. doi: 10.1093/ajcn/nqaa309. No abstract available. PMID 33301007
- [Derived] Martins C, Roekenes J, Hunter GR, Gower BA. Association between ketosis and metabolic adaptation at the level of resting metabolic rate. Clin Nutr. 2021 Aug;40(8):4824-4829. doi: 10.1016/j.clnu.2021.06.029. Epub 2021 Jul 6. PMID 34358822